CLINICAL TRIAL: NCT04670068
Title: A Phase 1 Study of Autologous Activated T-cells Targeting the B7-H3 Antigen in Subjects With Recurrent Epithelial Ovarian Cancer
Brief Title: Phase I Study of Autologous CAR T-Cells Targeting the B7-H3 Antigen in Recurrent Epithelial Ovarian
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC1818-ATL; R01CA256898 (NIH)
Record Dates: First submitted 2020-12-09; First posted 2020-12-17 (Actual); Results first posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Epithelial Ovarian Cancer
Keywords: Ovarian Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Ovarian Neoplasms | interventions — Immunotherapy, Adoptive; fludarabine; fludarabine phosphate; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CAR.B7-H3 T cell product (Experimental): Up to 12 patients will receive three weekly CAR.B7-H3 T cell product infusions at the same dose. To determine the recommended phase 2 dose (RP2D), a modified 3+3 dose escalation design will be used to evaluate two dose levels: Dose Level 1 (7.5x10^7 cells/infusion), Dose Level 2 (2x10^8 cells/infusion). If this dose is not tolerated, then a lower dose of 3.75 × 10^6 cells/infusion will be explored. Up to 3 dose levels of CAR.B7-H3 cells will be tested with at least 3 patients enrolled at each dose cohort before dose escalation is considered based on the incidence of dose limiting toxicity (DLT). An expansion cohort will enroll up to 9 patients at the recommended phase 2 dose. Prior to receiving the infusions, patients will undergo lymphodepletion with fludarabine and cyclophosphamide.
  Interventions: Drug: CAR.B7-H3; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: CAR.B7-H3 — Two dose levels will be evaluated: Dose Level 1 (7.5x10^7 cells/infusion), dose Level 2 (2x10^8 cells/infusion). If dose limiting toxicities (DLTs) are observed per protocol, Dose Level -1 (3.75x10^6 cells/infusion) will be evaluated.
  Other Names: Chimeric antigen receptor T cells with B7.H3 molecular target
Drug: Fludarabine — 30 mg/m^2 IV for 3 consecutive days
  Other Names: FLUDARA
Drug: Cyclophosphamide — 300 mg/m^2 IV for 3 consecutive days
  Other Names: Cytoxan

SUMMARY:
This is single center, open-label phase 1 dose escalation trial that uses modified 3+3 design to identify a recommended phase 2 dose (RP2D) of CAR.B7-H3 T cell product. An expansion cohort will enroll additional subjects at the RP2D for a total enrollment of up to 21 subjects on the protocol.

DETAILED DESCRIPTION:
This study is intended for the patients who have been diagnosed with Epithelial Ovarian Cancer that either came back or did not improve after previous treatments. The purpose of this study is to test the safety of using a new treatment called autologous T lymphocyte chimeric antigen receptor cells against the B7-H3 antigen (CAR.B7-H3 T cells) in patients with ovarian cancer. This treatment has not been approved by the Food and Drug Administration.

The study investigator's goal is to calculate the Maximum tolerated dose of the CAR.B7-H3 cells There are two parts to this study. In part 1, subject's blood sample will be used to manufacture the CAR.B7-H3 T cells.

Ovarian cancer cells carry a substance called B7-H3 which is not found in other healthy cells. the subject's T cells will be modified to make CAR.B7-H3 T cells so they may attack and destroy ovarian cancer cells that carry the B7-H3 substance. The CAR.B7-H3 T cells are given through a catheter in the abdomen, after completing three rounds of lymphodepletion chemotherapy. Lymphodepletion chemotherapy prepares the body to receive the CAR.B7-H3 T cells.

In part 2 of the study, the subjects will receive the CAR.B7-H3 T cells. Eligible patients will receive lymphodepletion chemotherapy with cyclophosphamide and fludarabine for three consecutive days. If they continue to meet the eligibility criteria, the modified CAR.B7-H3 T cells will be given to them 2-14 days after the last lymphodepletion chemotherapy session. Three infusions of the CAR.B7-H3 T cells may be given to the subject through a catheter in the abdomen. Infusions will be done once a week.

Lymphodepletion chemotherapy and infusion of the CAR.B7-H3 T cells will happen at UNC Cancer Hospital. On the days the subjects receive the CAR.B7-H3 T cells infusion- Blood, fluid, and tumor samples will be collected from the subject for research purposes. Tumor biopsies are a mandatory part of this research.

Post infusion visits are - 3, 4, and 6 weeks. Additional visits will happen every 3 months for one year after the last infusion. Similar follow-up clinic visits will be completed annually, for a total of 5 years.

This is a research study to obtain new information that may help people in the future.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for the Study

1. Written informed consent and HIPAA authorization for release of personal health information explained to, understood by, and signed by the subject or their legally authorized representative; subject was given a copy of the informed consent form.
2. Older than 18 years at the time of consent.
3. Subject has adequate performance status as defined by ECOG score of ≤ 2.
4. Subjects must have histologically or cytologically confirmed epithelial ovarian, peritoneal or fallopian tube cancer and must have a histological diagnosis of high-grade serous histology based on local histopathological findings.
5. Subjects must have recurrent platinum-resistant or platinum-refractory disease defined as:

   1. Disease that has progressed by imaging while receiving platinum OR
   2. Disease that has recurred within 6 months of the last receipt of platinum-based chemotherapy. Rising CA-125 only is not considered as a platinum-resistant or refractory disease.
   3. Having received at least 2 prior regimens.
   4. Have failed prior therapy with a PARP inhibitor if the subject has a germline or somatic BRCA mutation.
6. Subjects must have an evaluable disease - defined as:

   1. Measurable disease per RECIST 1.1 OR
   2. Non-measurable disease (defined as solid and/or cystic abnormalities on radiographic imaging that do not meet RECIST 1.1 definitions for target lesions) OR
   3. Ascites and/or pleural effusion that has been pathologically demonstrated to be disease-related in the setting of a CA-125 > 2 × ULN.

8. Subjects must be able to have an intraperitoneal port placed either by vascular interventional radiology or surgically in the operating room. (Note: The intraperitoneal port will not be placed until the subject is determined to be otherwise eligible to receive the CAR.B7-H3 infusion and until the subject is determined to be otherwise eligible to receive lymphodepletion).

9. Female subjects of childbearing potential must be willing to abstain from heterosexual activity or to use 2 forms of highly effective methods of contraception from the time of informed consent until 180 days after study treatment discontinuation. The two contraception methods can be comprised of two barrier methods, or a barrier method plus a hormonal method or an intrauterine device that meets < 1% failure rate for protection from pregnancy in the product label.

10. Subject is willing and able to comply with study procedures based on the judgment of the investigator or protocol designee.

11. Subject is willing to undergo a biopsy prior to treatment, at the time of final infusion, intraperitoneal catheter removal, and at the time of disease progression, and the tumor site is determined to be safe by the treating investigator for biopsy collection.

Eligibility Criteria Prior to Cell Procurement

1. Written informed consent to undergo cell procurement is explained to, understood by, and signed by the subject; the subject is given a copy of the informed consent form for cell procurement.
2. Subject has a life expectancy of≥ 3 months.
3. Subject has evidence of adequate organ function as defined by:

   1. Total bilirubin ≤ 1.5 × ULN, unless attributed to Gilbert's Syndrome
   2. AST / ALT ≤ 3 × ULN (Note: if intrahepatic liver metastases are present, AST and ALT must be ≤ 5 × ULN)
   3. Creatinine ≤ 2 × ULN
   4. Left ventricular ejection fraction (LVEF) • 40%, as measured by ECHO, with no additional evidence of decompensated heart failure.
4. Imaging results from within 90 days prior to procurement to assess the presence of active disease.
5. Female subjects of childbearing potential must have a negative serum pregnancy test within 72 hours prior to cell procurement. Note: Females are considered of childbearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months. Documentation of postmenopausal status must be provided.

Exclusion Criteria:

1. Subject is pregnant or lactating (Note: Breast milk cannot be stored for future use while the mother is being treated in the study).
2. Subject is deemed unlikely to be a candidate for successful intraperitoneal catheter placement by radiographic assessment.
3. Subject has intraparenchymal lung metastases (note that pleural effusions are not exclusionary and that subjects with intraparenchymal liver disease and subjects with the retroperitoneal disease are allowed on the study).
4. Subject has brain metastases. A subject with prior brain metastasis may be considered if they have completed their treatment for brain metastasis at least 4 weeks prior to being screened for eligibility, have been off of corticosteroids for ≥ 2 weeks, and are asymptomatic.
5. Subject has current signs and/or symptoms of bowel obstruction or signs and/or symptoms of bowel obstruction within 3 months prior to starting treatment.
6. Subject has a history of an intra-abdominal abscess within the past 3 months.
7. Subject has a history of gastrointestinal perforation.
8. The subject has a history of symptomatic diverticular disease, confirmed by CT or colonoscopy.
9. Subject is dependent on intravenous hydration or total parenteral nutrition.
10. Subject has a known additional malignancy that is active and/or progressive and requiring treatment; exceptions include basal cell or squamous cell skin cancer, in situ cervical or bladder cancer, or other cancer for which the subject has been disease-free for at least five years.
11. Current use of systemic corticosteroids at doses ≥10 mg prednisone daily or it's equivalent; those receiving <10 mg daily may be enrolled at the discretion of the investigator.
12. Subject has active infection with HIV, HTLV, HBV, and HCV (tests can be pending at the time of cell procurement; only those samples confirming lack of active infection will be used to generate transduced cells). Note: To meet eligibility subjects are required to be negative for HIV antibody or HIV viral load, negative for HTLV1 and 2 antibodies or PCR negative for HTLV1 and 2, negative for Hepatitis B surface antigen, negative for HCV antibody or HCV viral load.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2030-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Van Le, MD, Principal Investigator — UNC
Locations (1):
- Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Golubovskaya V. CAR-T Cells Targeting Immune Checkpoint Pathway Players. Front Biosci (Landmark Ed). 2022 Apr 2;27(4):121. doi: 10.31083/j.fbl2704121. PMID 35468680
- See also: Related Info — https://unclineberger.org/research/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants enrolled between 01/27/2021 - 12/19/2024 one center in North Carolina.
Groups:
- Arm 1 - Dose Level 1: Participants received Dose Level 1 (7.5x10^7 cells/infusion).
- Arm 2- Dose Level 2: Participants received Dose Level 2 (2x10^8 cells/infusion).
Period: Overall Study
Arm/Group | Arm 1 - Dose Level 1 | Arm 2- Dose Level 2
Started | 3 | 1
Completed | 1 | 0
Not Completed | 2 | 1
Not completed — Progressive Disease | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 2 - Dose Level 2: Participants received Dose Level 2 (2x10^8 cells/infusion).
- Total: Total of all reporting groups
Arm/Group | Arm 1 - Dose Level 1 | Arm 2 - Dose Level 2 | Total
Number analyzed (Participants) | 3 | 1 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 2
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs) Based on National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE)
Description: Dose-limiting toxicity (DLT) assessments will include toxicities that are at least possibly related to the CAR.B7-H3 T cell product and that occur from the day of the initial infusion through four weeks after the final administration. DLTs are defined as toxicities of Grade ≥3. All toxicities will be classified and graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE), version 5.0, which rates severity from Grade 1 (mild) to Grade 5 (death).
Time Frame: Up to 10 weeks (Up 4 weeks after the last CAR-T cell infusion)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 - Dose Level 1 | Arm 2- Dose Level 2
Number analyzed (Participants) | 3 | 1
Participants | 0 | 0

2. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs) Based on Cytokine Release Syndrome (CRS)
Description: Dose-limiting toxicities (DLTs) will include any toxicity that is at least possibly related to the CAR.B7-H3 T cell product and occurs from the first infusion through 4 weeks after the final dose. DLTs are defined as Grade ≥3 cytokine release syndrome (CRS) that does not improve to Grade ≤2 within 7 days. CRS will be graded per protocol criteria on a Grade 1 (mild) to Grade 5 (death) scale.
Time Frame: Up to 10 weeks (Up 4 weeks after the last CAR-T cell infusion)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 - Dose Level 1 | Arm 2- Dose Level 2
Number analyzed (Participants) | 3 | 1
Participants | 0 | 0

3. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs) Based on Immune Effector Cell-Associated Neurotoxicity Syndrome (ICANS)
Description: Dose-limiting toxicity (DLT) assessments will include any toxicity that is at least possibly related to the CAR.B7-H3 T cell product, occurring from the day of the first infusion through four weeks after the final cell product administration. DLTs are defined as Grade ≥3 Immune Effector Cell-Associated Neurotoxicity Syndrome (ICANS) or any other Grade ≥3 non-hematologic toxicity, including allergic reactions to T cell infusions. ICANS will be graded using protocol-defined criteria on a scale from Grade 1 (mild) to Grade 4 (critical). Cytokine Release Syndrome (CRS), if observed, will be graded on a scale from Grade 1 (mild) to Grade 5 (death), per the criteria outlined in the protocol.
Time Frame: Up to 10 weeks (Up 4 weeks after the last CAR-T cell infusion)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 - Dose Level 1 | Arm 2- Dose Level 2
Number analyzed (Participants) | 3 | 1
Participants | 0 | 0

4. Secondary Outcome: Disease Control Rate (DCR)
Description: Disease control rate will be defined as the percentage of subjects with complete response (CR), partial response (PR), and/or stable disease at 6 months per RECIST 1.1 criteria.
  Radiographic response will be measured by RECIST (Response Evaluation Criteria In Solid Tumors) Criteria, indicating if subject experienced a Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), no response or less response than Partial or Progressive; or Progressive Disease (PD), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 6 months after initial CAR-T cell infusion
Reporting Status: Not Posted

5. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression free survival (PFS) will be measured from the time of lymphodepletion prior to infusion with CAR.B7-H3 to progression (as defined per RECIST 1.1) or death.
  Radiographic response will be measured by RECIST, Response Evaluation Criteria In Solid Tumors Criteria, indicating if subject experienced a Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), no response or less response than Partial or Progressive; or Progressive Disease (PD), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From the date of lymphodepletion to the date of progression or death up to 5 years
Reporting Status: Not Posted

6. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) will be measured from the date of lymphodepletion prior to CAR.B7-H3 T cell product administration to the date of death.
Time Frame: From the date of lymphodepletion to the date of death up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 91 days
Description: Adverse events were monitored from procurement through the 4-week follow-up period after cellular treatment ended.
  All hospital admissions were considered Serious Adverse Event (SAE) per protocol.
Arm/Group | Arm 1 - Dose Level 1 | Arm 2- Dose Level 2
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/1
Other Adverse Events (participants affected / at risk) | 3/3 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 - Dose Level 1 (N=3) | Arm 2- Dose Level 2 (N=1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Cytokine release syndrome (Immune system disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 - Dose Level 1 (N=3) | Arm 2- Dose Level 2 (N=1)
Anemia (Blood and lymphatic system disorders) | 2 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Ascites (Gastrointestinal disorders) | 0 | 1
Bloating (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Edema limbs (General disorders) | 1 | 1
Fatigue (General disorders) | 3 | 1
Fever (General disorders) | 1 | 0
Generalized edema (General disorders) | 0 | 1
Pain (General disorders) | 1 | 1
Bruising (Injury, poisoning and procedural complications) | 0 | 1
Alkaline phosphatase increased (Investigations) | 1 | 1
lactate dehydrogenase increased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 3 | 1
Neutrophil count decreased (Investigations) | 3 | 1
Platelet count decreased (Investigations) | 1 | 0
White blood cell decreased (Investigations) | 3 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 2 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatremia (Metabolism and nutrition disorders) | 2 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1
Urinary tract pain (Renal and urinary disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0
Vaginal inflammation (Reproductive system and breast disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Hematoma (Vascular disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
This study was closed to accrual before reaching target accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-12): https://cdn.clinicaltrials.gov/large-docs/68/NCT04670068/Prot_SAP_000.pdf